CLINICAL TRIAL: NCT01902576
Title: Chronic GVHD Response Measures Validation
Status: Active, not recruiting | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2710.00; RG1000980 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples (30mL) processed for peripheral blood mononuclear cells (PBMC), plasma, and granulocytes.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to develop and validate endpoint measures that can accurately determine whether patients are responding to treatment for chronic Graft-versus-Host Disease (GVHD). Hopefully, this will also lead to being better able to predict which patients will respond to what therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 years or older
* Prior first allogeneic stem cell transplant, with any graft source, donor type, and GVHD prophylaxis.
* Diagnosis of chronic GVHD according to the criteria of the diagnosis and scoring group of the NIH consensus conference (Patient must have at least one diagnostic manifestation of chronic GVHD or one distinctive manifestation with pathological confirmation of the diagnosis. Concurrent acute GVHD manifestations will be allowed as long as at least one classic chronic manifestation is present.)
* Initiation of a new systemic treatment for chronic GVHD in the past 4 weeks or anticipated within the next 4 weeks. Systemic treatment is defined as any medication or intervention that has intended systemic effects, including extracorporeal photopheresis, regardless of prior lines of therapy or prior treatment with the agent(s). If a patient is restarting a treatment to which they were previously exposed, they must have been off of it for at least 4 weeks before restarting.
* No evidence of persistent or progressive malignancy at the time of enrollment
* Evaluation at the transplant center at the time of study enrollment, and agreement to be re-evaluated at the transplant center up to four subsequent times: at 3 months, 6 months, and 18 months after enrollment and once if another treatment is added for chronic GVHD.
* Signed, informed consent

Exclusion Criteria:

* Inability to comply with study procedures
* Complete resolution of chronic GVHD at the time of enrollment (patient must have some measurable chronic GVHD activity)

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients starting initial or subsequent therapy for chronic Graft vs Host Disease.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Develop and validate the Chronic GVHD-Activity Index (CGVHD-AI) as a measure of treatment response. | 18 months
  This measure is intended to capture impairments caused by chronic GVHD. We expect that change in the CGVHD-AI could be used to measure treatment response because it will correlate with clinically significant changes reported by physicians and patients. The CGVHD-AI would be most appropriate for use in clinical trials where the goal is symptom relief and decreased disease activity.

SECONDARY OUTCOMES:
To develop and validate the Chronic GVHD Failure-Free Survival Score (CGVHD-FFS) as a predictor of failure-free survival. | 18 months
  This measure is intended for use as an intermediate endpoint that predicts subsequent failure-free survival, defined as absence of death, relapse and requirement for new therapy, i.e., events that constitute treatment failures in clinical trials. The CGVHD-FFS would be most appropriate for phase II and III trials testing agents intended to change the underlying biology of the syndrome, for example by inducing immunologic tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Lee, MD MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Inamoto Y, Martin PJ, Onstad LE, Cheng GS, Williams KM, Pusic I, Ho VT, Arora M, Pidala J, Flowers MED, Gooley TA, Lawler RL, Hansen JA, Lee SJ. Relevance of Plasma Matrix Metalloproteinase-9 for Bronchiolitis Obliterans Syndrome after Allogeneic Hematopoietic Cell Transplantation. Transplant Cell Ther. 2021 Sep;27(9):759.e1-759.e8. doi: 10.1016/j.jtct.2021.06.006. Epub 2021 Jun 12. PMID 34126278